CLINICAL TRIAL: NCT07392554
Title: Virtual Reality as a Tool for Training Public Speaking Skills in Higher Education Students: A Randomized Controlled Trial
Brief Title: Virtual Reality as a Tool for Training Public Speaking Skills in Higher Education Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Fonds pour la Recherche Scientifique (FRS-FNRS) (Unknown)
Responsible Party: Principal Investigator, Lamia BETTAHI, PhD Student, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CE 2526-003 - FRESH FC 52277
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Voice; Speech; Virtual Reality Simulation; Healthy Adult
Keywords: Public Speaking; Oral Communication; Voice; Speech Fluency; Speech Therapy; Virtual Reality; Students; Training; Glossophobia; Anxiety; Verbal Behavior
MeSH Terms: conditions — Speech; Communication Disorders; Glossophobia; Anxiety Disorders; Verbal Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): * Indirect method: one information session on general advice about PS
  * Direct method: three sessions of PS training including VR simulations over a course of 3 weeks.
  Interventions: Behavioral: Indirect Method; Behavioral: Direct Method
- Wait-list control arm (Other): * Indirect method: one information session on general advice about PS
  * Delayed direct method: after a waiting period of three weeks, three sessions of PS training including simulations over a course of 3 weeks.
  Interventions: Behavioral: Indirect Method; Behavioral: Direct Method

INTERVENTIONS:
Behavioral: Indirect Method — • General information and advice on PS
Behavioral: Direct Method — • Learning effective PS oral skills using speech therapy exercises (e.g., modeling, audiovisual feedback) and VR simulations

SUMMARY:
According to the scientific literature, public speaking (PS) is an important skill for students to master. However, a large proportion of students do not feel comfortable speaking in public. PS anxiety impacts oral communication (i.e., voice and fluency). These changes can affect speaker's academic and professional success, as well as his credibility. Performing a high-quality PPP with confidence is therefore rarely an innate skill, but fortunately it can be trained and improved. Therefore, training PS skills in representative settings is crucial but often challenging for PS professionals (e.g., speech therapists, vocologists, coaches).

This project examines how oral communication skills training including simulations in virtual reality (VR) supports the acquisition of effective oral PS skills. Using acoustic analyses, outcomes from participants in the intervention group (N = 40) will be compared with those of a wait-list control group (N = 40) to determine whether significant differences emerge in filled pauses, speech rate, and vocal intonation during PS. Changes in PS self-efficacy will also be assessed. Regarding secondary outcomes, the study will evaluate changes in self-reported and physiological PS anxiety, as well as self-reported confidence as a speaker. Finally, self-perceived vocal effort during PS will be examined.

DETAILED DESCRIPTION:
The present study is a randomized wait-list control trial, i.e. participants are randomly assigned to either the group that receives the intervention directly or the group that receives the intervention after a waiting period. First, both groups will receive a 1-hour session of information on general advice about PS (indirect method). Then the participants in the experimental group will receive three 1-hour sessions of voice and fluency training with VR practice moments for a period of 3 weeks (direct method). The control wait-list group will first wait for 3 weeks and then get the direct method training. The investigators will collect data from all participants in the first week (before the start of intervention for the experimental group), fourth week (right after the intervention for the experimental group and right before the first intervention session for the control group) and seventh week (three weeks after the intervention for the experimental group and right after the intervention for the control group).

ELIGIBILITY:
Inclusion Criteria:

* Higher education student
* Speaking french fluently

Exclusion Criteria:

* Hearing impairment
* Voice or fluency disorder at the time of the study

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Filled pauses | Week 1(baseline), 4 and 7
  Measurements of participants' filled pauses (percentage of the total number of syllables produced) when PS in VR
Speech rate | Week 1(baseline), 4 and 7
  Measurements of participants' speech rate (in syllables per second) when PS in VR
Voice intonation | Week 1(baseline), 4 and 7
  Acoustic measurements of participants' voice variation (in semitones) when PS in VR
PS self-efficacy | Week 1(baseline), 4 and 7
  Questionnaire on self-efficacy in PS

SECONDARY OUTCOMES:
Self-reported PS anxiety | Week 1(baseline), 4 and 7
  Self-assessment of perceived anxiety using the Subjective Units of Distress Scale (SUDS)
Physiological PS anxiety | Week 1(baseline), 4 and 7
  Measurements of participants' heart rate (in bpm) when PS in VR
Self-reported confidence as a speaker | Week 1(baseline), 4 and 7
  Self-assessment of confidence as a speaker using the Personal Report of Confidence as a Speaker (PRCS) short-form questionnaire
Self-perceived vocal effort | Week 1(baseline), 4 and 7
  Self-assessment of perceived vocal effort using the Adapted BORG Category Ratio (CR-10) physical exertion scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No